CLINICAL TRIAL: NCT04963296
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study To Evaluate The Efficacy And Safety of Obinutuzumab in Patients With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Efficacy and Safety of Obinutuzumab in Participants With Systemic Lupus Erythematosus
Acronym: ALLEGORY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA42750; 2020-005760-57 (EudraCT Number); 2023-504774-38-00 (Other: EU CT Number)
Record Dates: First submitted 2021-07-07; First posted 2021-07-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — obinutuzumab; Acetaminophen; Diphenhydramine; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obinutuzumab (Experimental): Participants will receive obinutuzumab 1000 milligrams (mg) intravenous (IV) infusions on Day 1 and at Weeks 2, 24 and 26.
  Interventions: Drug: Obinutuzumab; Drug: Acetaminophen/Paracetamol; Drug: Diphenhydramine hydrochloride; Drug: Methylprednisolone
- Placebo (Placebo Comparator): Placebo participants will receive obinutuzumab matched placebo on Day 1 and at Weeks 2, 24 and 26.
  Interventions: Drug: Placebo; Drug: Acetaminophen/Paracetamol; Drug: Diphenhydramine hydrochloride; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab will be administered by IV infusion at a dose of 1000 mg on Day 1 and at Weeks 2, 24 and 26.
  Other Names: Gazyva, GA101, RO5072759
  Arms: Obinutuzumab
Drug: Placebo — Placebo matching obinutuzumab will be administered by IV on Day 1 and at Weeks 2, 24 and 26.
  Arms: Placebo
Drug: Acetaminophen/Paracetamol — Acetaminophen 650-1000 mg will be administered as premedication prior to infusions.
Drug: Diphenhydramine hydrochloride — Diphenhydramine 50 mg will be administered as premedication prior to infusions.
Drug: Methylprednisolone — Methylprednisolone 80 mg IV will be administered as premedication prior to infusions.

SUMMARY:
This parallel-group, double-blind, placebo-controlled study will evaluate the efficacy and safety of obinutuzumab versus placebo in participants with active, autoantibody-positive systemic lupus erythematosus (SLE) who are treated with standard-of-care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) Classification Criteria >=12 weeks prior to screening
* Anti-nuclear antibody (ANA) >=1:80, or anti-dsDNA and/or anti-Sm antibodies above the upper limit of normal (ULN), as determined by the central laboratory at screening
* Low C3 or low C4 or low CH50 complement as determined by the central laboratory at screening
* High disease activity at screening, based on; BILAG-2004 (Category A disease in >=1 organ system and/or Category B disease in >=2 organ systems), Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) (score >=8) and Physician's Global Assessment (PGA) (score >=1.0 on a 0 to 3 visual analogue scale [VAS])
* High disease activity on Day 1, based on; SLEDAI-2K (score >=8) and PGA (score >=1.0 on a 0 to 3 VAS)
* Current receipt of >=1 of the following classes of standard therapies for the treatment of SLE at stable doses: oral corticosteroid (OCS), antimalarials, conventional immunosuppressants
* Other inclusion criteria may apply
* The Medical Monitor may be consulted if there are any questions related to eligibility criteria

Exclusion Criteria:

* Pregnancy or breastfeeding
* Presence of significant lupus-associated renal disease and/or renal impairment
* Receipt of an excluded therapy, including any anti-CD20, anti-CD19 therapy less than 9 months prior to screening or during screening; or cyclophosphamide, tacrolimus, ciclosporin, or voclosporin during the 2 months prior to screening or during screening
* Significant or uncontrolled medical disease which, in the investigator's opinion, would preclude patient participation
* Known active infection of any kind or recent major episode of infection
* Intolerance or contraindication to study therapies
* Other exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2028-03-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Systemic Lupus Erythematosus Responder Index (SRI[4]) at Week 52 | Week 52
  SRI(4) requires reduction from baseline of >=4 points in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K), no new systems or organs affected, as defined by >=1 new British Isles Lupus Assessment Group (BILAG) A or >=2 new BILAG B items compared with baseline using BILAG-2004, and no worsening from baseline of >=0.30 points on a 3-point Physician's Global Assessment Visual Analogue Scale (PGA-VAS).

SECONDARY OUTCOMES:
Percentage of Participants who Achieve SRI(6) at Week 52 | Week 52
  SRI(6) requires reduction from baseline of >=6 points in the SLEDAI-2K, no new systems or organs affected, as defined by >=1 new BILAG A or >=2 new BILAG B items compared with baseline using BILAG-2004, and no worsening from baseline of >=0.30 points on a 3-point PGA-VAS.
Percentage of Participants Entering the Study on Prednisone >= 10 mg/day (or equivalent) who Achieve Sustained Corticosteroid Control | From Week 40 to Week 52
  No treatment with prednisone >=7.5 mg/day (or equivalent) and no receipt of intravenous, intramuscular, or intra-articular corticosteroids.
Time to First BILAG Flare over 52 Weeks | From baseline to Week 52
  Flare is defined as the occurrence of >=1 new BILAG A or >=2 new BILAG B manifestations from the previous visit
Percentage of Participants who Achieve a Sustained SRI(4) Response | From Week 40 to Week 52
  Achievement of SRI(4) at all study visits from Week 40 through Week 52.
Percentage of Participants who Achieve British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) at Week 52 | Week 52
  Reduction of all baseline BILAG-2004 A items to B/C/D and baseline BILAG-2004 B items to C/D; no new systems or organs affected, as defined by >=1 new BILAG A or >=2 new BILAG B items compared with baseline; no net increase in SLEDAI-2K score from baseline; and no worsening from baseline of >=0.30 points on a 3-point PGA-VAS.
Percentage of Participants who Achieve SRI(8) at Week 52 | Week 52
Percentage of Participants who Achieve SRI(4) at Week 24 | Week 24
Percentage of Participants who Achieve Clinical SRI(4) at Week 52 | Week 52
Percentage of Participants who Achieve SRI(4) at Week 52 on Low-dose Corticosteroids | Week 52
Percentage of Participants who Achieve Lupus Low Disease Activity State (LLDAS) at Week 52 | Week 52
Percentage of Participants who Achieve Definition of Remission in SLE (DORIS) at Week 52 | Week 52
Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale | From baseline to Week 24 and from baseline to Week 52
Change in 36-Item Short Form Survey, Version 2 (SF-36 v2) Bodily Pain Domain Scale | From baseline to Week 24 and from baseline to Week 52
Change in SF-36 v2 Physical Component Summary Scale | From baseline to Week 24 and from baseline to Week 52
Change in Active Joint Count (Swollen plus Tender) | From baseline to Week 24 and from baseline to Week 52
Percentage of Participants who Achieve a >= 50% Reduction in Active Joint Counts (Swollen plus Tender) at Each Study Visit | From baseline to Week 52
Percentage of Participants who Achieve a >= 50% Reduction in Cutaneous Lupus Erythematosus Disease Area and Severity (CLASI) Total Activity Score at each Study Visit, among Participants with CLASI Total Activity Score >=10 at Baseline | From baseline to Week 52
Percentage of Participants who Achieve Sustained Corticosteroid Control | From Week 40 through Week 52
Cumulative Corticosteroid use (in Equivalent Milligrams of Prednisone) | From baseline to Week 52
Annualized flare rate through Week 52 | At Week 52
Percentage of Participants with Adverse Events | From baseline to approximately 6 years
Percentage of Participants with Adverse Events of Special Interest (AESIs) | From baseline to approximately 6 years
Serum Concentration of Obinutuzumab | Double blind period: At Weeks 2, 4, 12, 24, 26, 36, 52 and at early study discontinuation visit; Open label period: At Weeks 54, 56, 58, 66, 78, 90, 104 and at early study discontinuation visit
Percentage of Participants with Anti-drug Antibodies (ADAs) at Baseline | Baseline
Percentage of Participants with ADAs During the Study | Up to approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (64):
- United States (14):
  - Pinnacle Research Group, Anniston, Alabama
  - Unity Health - White County Medical Center- Rheumatology, Searcy, Arkansas
  - Providence Medical Foundation, Fullerton, California
  - Arthritis & Rheumatism, Aventura, Florida
  - Great Lakes Center of Rheumatology, Lansing, Michigan
  - Clinical Research Institute of Michigan, LLC, Troy, Michigan
  - Northwell Health Division of Rheumatology, Great Neck, New York
  - Columbia University Medical Center, New York, New York
  - Joint & Muscle Research Institute, Charlotte, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Texas Arthritis Center, El Paso, Texas
  - Prolato Clinical Research Center, Houston, Texas
- Argentina (3):
  - Organizacion Medica de Investigacion, Buenos Aires
  - DOM Centro de Reumatología, Buenos Aires
  - Centro de Investigaciones Médicas Tucuman, San Miguel
- Brazil (7):
  - Ser Servicos Especializados Em Reumatologia, Salvador, Estado de Bahia
  - Hospital das Clinicas - UFMG, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericordia, Belo Horizonte, Minas Gerais
  - Centro Mineiro de Pesquisa - CMIP, Juiz de Fora, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras ? CETI, Curtiba, Paraná
  - Hospital das Clinicas - FMUSP Ribeirao Preto, Ribeirão Preto, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos - CEMEC*X*, São Bernardo do Campo, São Paulo
- Revmatologicky Ustav, Prague, Czechia
- Ch Pitie Salpetriere, Paris, France
- Italy (5):
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - IRCCS S. Raffaele, Milan, Lombardy
  - A.O. Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliero-Universitaria Di Ferrara Arcispedale Santanna, Cona (Ferrara), Veneto
  - Uni Di Padova, Padua, Veneto
- Mexico (5):
  - Centro de Investigacion Alberto Bazzoni S.A. de C.V., Torreón, Coahuila
  - Unidad de Reumatologia Rehabilitacion Integral, Mexicali, Estado de Baja California
  - Centro de Investigación y Tratamiento Reumatológico S.C., Mexico City, Mexico CITY (federal District)
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro de Investigación de Tratamientos Innovadores de Sinaloa (CITI), Culiacán, Sinaloa
- New Zealand (2):
  - Middlemore Hospital, Auckland
  - Wellington Hospital, Wellington
- Peru (5):
  - Hogar Clínica San Juan de Dios, Arequipa
  - Clínica San Juan Bautista CSJB, Lima
  - Instituto de Ginecología y Reproducción, Lima
  - Clinica El Golf, San Isidro
  - Clinica San Antonio;Investigaciones Trujillo S.A.C., Trujillo
- Poland (7):
  - Szpital Uniwersytecki, Bydgoszcz
  - Medyczne Centrum Hetmanska, Poznan
  - Prywatna Praktyka Lekarska, Poznan
  - Ortopedyczno Rehab Szpital Klinic im Wiktora Degi UM, Poznan
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - REUMATOP Grzegorz Rozumek, Karin Pistorius Spó?ka Jawna, Wroc?aw
- Russia (3):
  - Republican clinical hospital named after G.G. Kuvatov, Ufa, Bashkortostan Republic
  - Federal State Budgetary Scientific Institution Research Institute of Rheumatology V.A. Nasonova, Moscow, Moscow Oblast
  - FGBU ?Federal Medical and Research Center named after V.A.Almazov? Russian Ministry of Health, Saint Petersburg, Sankt-Peterburg
- South Africa (4):
  - Panorama Medical Center, Cape Town
  - Winelands Medical Research, Cape Town
  - Emmed Research, Pretoria
  - Dr Asokan Naidoo, Umhlanga
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
- United Kingdom (5):
  - Addenbrooke'S Hospital, Cambridge
  - Chapel Allerton Hospital, Leeds
  - Royal Free Hospital, London
  - Guy's Hospital, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing